CLINICAL TRIAL: NCT01838707
Title: Postoperative Epidural Analgesia in Spine Fusion Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omnia Askar, assistant lecturer of anesthesia and ICU, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1976
Record Dates: First submitted 2013-04-20; First posted 2013-04-24 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Pain
Keywords: postoperative; spine surgery
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (3):
- Bupivacaine (Active Comparator): 0.125% Bupivacaine HCL @ 4-5 ml/h
  Interventions: Drug: 0.125% Bupivacaine HCL @ 4-5 ml/h
- Bupivacaine, Morphine (Active Comparator): 0.125% Bupivacaine HCL , Morphine sulphate 3 mg @ 3-5 ml/h
  Interventions: Drug: 0.125% Bupivacaine HCL , Morphine sulphate @ 3 mg 3-5 ml/h
- Bupivacaine, Fentanyl (Active Comparator): 0.125% Bupivacaine, Fentanyl 100 mic @ 3-5 ml/h
  Interventions: Drug: 0.125% Bupivacaine, Fentanyl 100 mic @ 3-5 ml/h

INTERVENTIONS:
Drug: 0.125% Bupivacaine HCL @ 4-5 ml/h
  Arms: Bupivacaine
Drug: 0.125% Bupivacaine HCL , Morphine sulphate @ 3 mg 3-5 ml/h
  Arms: Bupivacaine, Morphine
Drug: 0.125% Bupivacaine, Fentanyl 100 mic @ 3-5 ml/h
  Arms: Bupivacaine, Fentanyl

SUMMARY:
we aim to compare the analgesic effect of 0.125% bupivacaine HCL, 0.125% bupivacaine HCL + Morphine sulphate 3 mg, 0.125% bupivacaine HCL + Fentanyl 100 micro gram both at rest and mobilization maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing spine fusion surgery.

Exclusion Criteria:

* Drug addiction. Intraoperative dural tear. Uses of opioids drug for any reason in the previous 48 hours. Mental dysfunction. Spinal fusion for any infectious or malignant causes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Assessment of pain | first 3 postoperative days
  • Pain will be assessed using the VAS ranging from "0" (no pain) to "10" (worst imaginable pain). Pain will be evaluated at rest, while coughing, and during mobilization. Maneuvers of particular clinical importance for postoperative mobilization (alone and with help) will be chosen: Turning in bed, standing in front of the bed and walking, and using the toilet without help. The time needed until the patient can first successfully perform these maneuvers will be documented.

SECONDARY OUTCOMES:
assessment of patients' satisfaction | First 3 postoperative days
  verbal rating score will be used (4 = very satisfied, 3 = satisfied, 2 = neutral, 1 = dissatisfied, and 0 = very dissatisfied).

OTHER OUTCOMES:
beta-endorphin | 1st postoperative day
  3 serum samples for beta-endorphin will be taken 1st one preoperative base line , 2nd at VAS more than 3 at rest ,3rd when VAS less than 2 at rest

CONTACTS AND LOCATIONS:
Overall Officials: Omnia A Abd El Raof, M.Sc., Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt